CLINICAL TRIAL: NCT01331967
Title: The Effect of Pioglitazone on Neointima Volume and Characteristics Observed by Optical Coherence Tomography (OCT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Associate professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRAISE II
Record Dates: First submitted 2011-04-05; First posted 2011-04-08 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Stable Angina; Diabetic Unstable Angina
Keywords: pioglitazone; optical coherence tomography; microRNA; neointima; major adverse cardiovascular event
MeSH Terms: conditions — Neointima | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Pioglitazone, Placebo (Experimental)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 15-30mg, once daily for 9 months

SUMMARY:
Pioglitazone is used in the treatment of diabetic patients. Thiazolidinediones increase insulin sensitivity and show favorable effect on blood glucose levels and lipid profiles. The effect of pioglitazone on atherosclerotic and inflammatory markers has not been compared in prospective manner after everolimus-eluting stent implantation by OCT. The purpose of this prospective, randomized, open-label trial is to compare the effect of pioglitazone on neointima volume and atherosclerosis progression in type 2 diabetic patients by using OCT. Moreover, changes in neointima characteristics could be analyzed along with the changes in miRNA-21, -126, -143, -145. Major adverse cardiovascular events such as non-fatal MI, death, stroke, and TLR could be compared.

DETAILED DESCRIPTION:
People with diabetes mellitus are more prone to coronary heart disease, stroke, and peripheral vascular disease, and diabetes mellitus has been regarded as an independent risk factor for the progression of coronary artery disease. Several studies have been reported that diabetes increased the risk of cardiovascular mortality in both men and women. With the introduction of drug-eluting stents (DESs), the angiographic rates of restenosis at later months have reduced dramatically in several studies. However, even with DESs, diabetic patients showed increased rates of restenosis and late loss index compared with nondiabetic patients. Diabetes has been considered to be a predictor of poor prognosis after percutaneous coronary intervention with drug-eluting stents. Long-term clinical and angiographic outcomes after percutaneous coronary intervention (PCI) with drug-metal stents (DESs) have been demonstrated to be worse in diabetic patients compared with nondiabetic patients. In the era of DESs, no study has demonstrated the clinical and angiographic outcomes in diabetic patients after DES implantation by using optical coherence tomography (OCT).

Various microRNAs such as miRNA-21, -126, -143, -145 are involved in the restenosis and atherosclerosis progression (Figure 1). Changes in these miRNAs from baseline to 9 months after randomization have never been studied, and the effects of pioglitazone in correlation with the changes in various miRNAs could be utilized in clinical practices. Comparison of pioglitazone and placebo on 9 months follow-up neointima volume and neointima characteristics by optical coherence tomography (OCT) will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* Gender eligible for study: both
* Diabetic patients either previously diagnosed or newly found diabetes.
* Fasting blood glucose ≥ 126 mg/dl or PP2 blood glucose ≥ 200 mg/dl for newly found diabetes.
* Patients with significant coronary artery disease (diameter stenosis > 70%) requiring stent implantation.
* Patients with informed consent.

Exclusion Criteria:

* Diabetic patients with the use of thiazolidinediones
* ACE inhibitor or ARB not allowed during the study period
* Previous history of PCI or bypass surgery
* Patients with any contraindications to the treatment of thiazolidinediones
* Pregnant or lactating patients
* Chronic alcohol or drug abuse
* Hepatic dysfunction
* Renal dysfunction
* Heart failure (EF < 50%)
* Expected life expectancy of < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
9 months follow-up neointima volume and neointima characteristics | 9 months follow-up
  Comparison of pioglitazone and placebo on 9 months follow-up neointima volume and neointima characteristics by optical coherence tomography (OCT). Moreover, changes in miRNA-21.-126, -143, -145 from baseline to 9 months will be compared.

SECONDARY OUTCOMES:
major adverse cardiovascular events | 9 months follow-up
  Comparison of pioglitazone and placebo on 9 months follow-up atheroma characteristics. Moreover, major adverse cardiovascular events such as non-fatal MI, death, stroke, and TLR will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea